CLINICAL TRIAL: NCT01638806
Title: Acute Versus Subacute Angioplasty in Patients With NON-ST-Elevation Myocardial Infarction (NON-ST-Elevation Myocardial Infarction=NONSTEMI Trial)
Brief Title: Acute Versus Subacute Angioplasty in Patients With NON-ST-Elevation Myocardial Infarction
Acronym: NONSTEMI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow recuritment
Sponsor: Aarhus University Hospital Skejby (Other)
Responsible Party: Principal Investigator, Christian Juhl Terkelsen, Associate professor, MD, PhD, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NONSTEMI
Record Dates: First submitted 2012-06-28; First posted 2012-07-12 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Myocardial Infarction
Keywords: Acute Coronary Syndrome; Myocardial infarction; Angioplasty; Prehospital emergency care; Biological markers; Troponin; Point-of-Care systems
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I: PPCI (Experimental): Patients are treated with Aspirin, ADP-blocker and heparin and field-triaged or transferred immediately to an invasive center for PPCI
  Interventions: Procedure: Group I: Primary PCI
- Conventional: Group II (No Intervention): Patients are treated as today: Admission to local hospital, Low-molecular-weight heparin (LMWH), Aspirin, ADP-blocker and within 72 hours transfer for angiography/angioplasty. Patients with a Grace score > 140 will be transferred for angiography/angioplasty within 24 hours. Patients with refractory angina, severe heart failure, life-threatening ventricular arrhythmias or haemodynamic instability will be transferred acutely for angiography/angioplasty according to the european guidelines.

INTERVENTIONS:
Procedure: Group I: Primary PCI — Patients are treated with Aspirin, ADP-blocker and heparin and field-triaged or transferred immediately to an invasive center for PPCI
  Other Names: PPCI in NONSTEMI
  Arms: Group I: PPCI

SUMMARY:
Patients with acute myocardial infarction (AMI) are categorized according to the electrocardiogram (ECG) findings into: 1) patients with ST-Elevation Myocardial Infarction (STEMI), 2) patients with Bundle Branch Block Myocardial Infarction (BBBMI), and 3) remaining patients with so-called NON-ST-Elevation Myocardial Infarction (NONSTEMI).

Patients with STEMI or BBBMI are treated with acute angioplasty (PPCI=primary percutaneous coronary intervention), and the sooner PPCI is performed the lower is the mortality. This is why prehospital diagnosis and field-triage of patients with STEMI directly to heart centers with PPCI facilities is recommended.

In patients with NONSTEMI previous trials have indicated that early angioplasty, within 72 hours of symptom onset, is associated with improved outcome when compared to late angioplasty or conservative therapy. No trials have so far been able to diagnose patients with NONSTEMI in the prehospital phase or immediately on arrival at a hospital, and triage them directly to PPCI. Implementation of point-of-care (POC) testing of biomarkers may enable prehospital or early inhospital establishment of the diagnosis NONSTEMI.

The aim of the present trial is to identify patients with NONSTEMI in the prehospital phase or immediately on arrival at the local hospital based on a) symptoms, b) POC testing and c) ECG findings and then randomize patients to I) PPCI, or II) medical therapy and angiography/angioplasty within 72 hours (todays routine).

Se below for detailed description

DETAILED DESCRIPTION:
In the present trial patients with a) typical angina pectoris (AP) combined with b1) rise in biomarkers on POC testing (prehospital/immediately inhospital) and/or b2) ST-segment depression of more than 0.2 mV in two contiguous leads or more than 0.1 mV in four contiguous leads are randomized to I) PPCI (same protocol as in STEMI patients) or II) medical therapy and angiography/angioplasty within 72 hours (todays routine practice).

The primary purposes of the present trial is threefold:

1. To evaluate if it is possible to diagnose patients with NONSTEMI in the prehospital phase or immediately on arrival at the hospital (N=250 patients)
2. To compare a combined endpoint of mortality, re-infarction (during index admission or readmitted), or readmission with Congestive Heart Failure (CHF) between group I (PPCI strategy) and group II (routine strategy) (N=2500 patients).
3. To compare mortality between group I and II (N=4500 patients).

Secondary purposes of the present trial is:

1. To evaluate whether there is difference in the primary endpoints in patients randomized within or after 12 hours of symptom onset.
2. To evaluate whether there is difference in the primary endpoints in patients randomized in the prehospital phase and on admission to the hospital, respectively.
3. To evaluate whether there is difference in the primary endpoints in patients with a final diagnosis of AMI, as adjudicated by a clinical event committee.
4. To evaluate whether there is difference in the primary endpoints in patients with or without diabetes, respectively.
5. To compare a combined endpoint of mortality, readmission with AMI, readmission with CHF, readmission with AP, revascularization (not planned on index admission).
6. To compare a combined safety endpoint of stroke or serious bleeding between group I and II.
7. To evaluate if there is difference in the frequency of PCI and CABG in group I versus II.
8. To compare total admission time between group I and II.
9. To compare total cost between group I and II.
10. To compare total duration where the patient is on sick leave between group I and II

ELIGIBILITY:
Inclusion Criteria:

* Angina
* Elevated biomarkers (Point-of-care testing) either prehospital or immediately on admission
* ST-segment depression of 0.2mV or more in two contiguous leads or 0.1 mV or more in four contiguous leads.
* Patient can be randomized either in the prehospital phase or within 30 minutes of admission to a hospital

Exclusion Criteria:

* Tachycardia > 120
* Age < 18 or > 80 years
* Indication for PPCI already fulfilled
* Dementia
* Patient cannot understand the study information
* Presumed "troponisme"
* Left ventricular hypertrophy
* Known dialysis
* Previous CABG
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2012-06; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Mortality | within 1 year from randomization
  all-cause mortality
Re-infarction | within 1 year from randomization
  Re-infarction (during index admission or readmitted) adjudicated by and endpoint committee. The endpoint committee is blinded to the initial randomization. The "Universal definition of Myocadial infarction" will be used to classify reinfarction. Biomarkers will be recorded with emphasis on the need of obtaining blood samples until a peak has been reached during index hospitaltization before reinfarction can be considered. Re-infarction will require a 20% relative rise in biomarker level.
Readmission with CHF | within 1 year from randomization
  Readmission or visit in the outpatient clinic with CHF. Readmission or visit with CHF needs to be adjudicated by an endpoint committee blinded to the initial randomization.
Confirmed AMI | during index admission
  An endpoint committee needs to evaluate whether each patient had AMI on the index admission. This evaluation is performed without the endpoint committee being aware whether the patient was randomized to PPCI or conventional therapy. The endpoint committee will classify whether the patient had: a) NONSTEMI, b) STEMI with symptom duration <=12 hours, c) STEMI with symptom duration >12 hours, d) BBBMI with symptom duration <=12 hours or e) BBBMI with symptom duration > 12 hours.

SECONDARY OUTCOMES:
Readmission with AP | within 3 months, 1 year, and 5 year from randomization
  The national health registry is used to determine whether the patient is readmitted with AP. Time from index admission to first readmission with AP is determined. The endpoint committee adjudicate readmissions with AP blinded to original treatment strategy (Group I versus II)
Readmission with stroke | within 3 months, 1 year, and 5 year from randomization
  The national health registry used to determine whether the patient is readmitted with stroke. Stroke was defined as focal loss of neurologic function caused by an ischemic or hemorrhagic event, with residual symptoms lasting at least 24 hours or leading to death. Time from index admission to first readmission with stroke is determined. The endpoint committee adjudicate readmissions with stroke blinded to original treatment strategy (Group I versus II).
Non-scheduled re-intervention | within 3 months, 1 year, and 5 year from randomization
  The national health registry is used to determine whether the patient has non-scheduled re-intervention performed (re-intervention not scheduled at index admission). Time from index admission to first re-intervention and type of re-interverntion (PCI or CABG) is determined. The endpoint committee adjudicate re-interventions blinded to original treatment strategy (Group I versus II)
Duration of index admission | Time from initial admission to discharge
  The national health registry is used to determine number of days the patietns was admitted during index hospitalization (local hospital and interventional hospital).
Sick-leave from work | within 3 months, 1 year, and 5 year from randomization
  The national DREAM database is used to determined whether the patient is on sick leave from work after index hospitalization and the duration of sick leave from work.
Total cost | within 3 months, 1 year, and 5 year from randomization
  The total cost for each treatment strategy is calculated: EMS-transport, admission, cost for PCI / CABG.
Bleeding | within 3 months, 1 year, and 5 year from randomization
  The national health registry is used to determine bleeding events. The same criteria for bleeding classification is used as in the PLATO trial (see NEJM 2009 for details) to categorize: 1) Major life-threatening bleeding, 2) Other major bleeding. In addition BARC type 4 (CABG-related) bleedings are registered.
Time to intervention | Time from ambulance call to PCI or CABG is performed or angiography is performed without indication for PCI or CABG
  The time frame is equal to the health care system delay (time from EMS call to intervention)
Cardiovascular mortality | within 3 months, 1 year, and 5 year from randomization
  Cardiovascular mortality according to the Danish Registry of Cause of Death.

CONTACTS AND LOCATIONS:
Overall Officials: Christian J Terkelsen, MD,PhD, Principal Investigator — Department of cardiology B, Aarhus University Hospital in Skejby, Denmark; Hans E Bøtker, MD,DmSc,Prof, Study Director — Department of cardiology B, Aarhus University Hospital in Skejby, Denmark; Carsten Stengaard, MD, Study Chair — Department of cardiology B, Aarhus University Hospital in Skejby, Denmark; Jacob T Sørensen, MD, PhD, Study Chair — Department of cardiology B, Aarhus Unversity Hospital in Skejby, Denmark
Locations (1):
- Department of cardiology, Aarhus University Hospital in Skejby, Aarhus, Denmark

REFERENCES:
- [Derived] Rasmussen MB, Stengaard C, Sorensen JT, Riddervold IS, Sondergaard HM, Niemann T, Dodt KK, Frost L, Jensen T, Raungaard B, Hansen TM, Giebner M, Rasmussen CH, Botker HE, Kristensen SD, Maeng M, Christiansen EH, Terkelsen CJ. Comparison of Acute Versus Subacute Coronary Angiography in Patients With NON-ST-Elevation Myocardial Infarction (from the NONSTEMI Trial). Am J Cardiol. 2019 Sep 15;124(6):825-832. doi: 10.1016/j.amjcard.2019.06.007. Epub 2019 Jun 24. PMID 31324357